CLINICAL TRIAL: NCT05121844
Title: Use of Continuous Glucose Monitoring in Non-Diabetic Population to Compliment Signos Mobile Health Platform: Comprehensive Weight Optimization Program and Customized Lifestyle Modifications
Brief Title: Use of Continuous Glucose Monitoring in Non-Diabetic Population to Compliment Signos Mobile Health Platform
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Signos Inc (Industry)
Responsible Party: Principal Investigator, Stephanie Kim, M.D., MPH, Principal Investigator, Signos Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 195165
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Weight Loss; Metabolic Syndrome; Pre-diabetes; Central Obesity; Glucose Intolerance; Metabolic Glucose Disorders
Keywords: health and wellness; excess adiposity
MeSH Terms: conditions — Weight Loss; Metabolic Syndrome; Glucose Intolerance; Obesity, Abdominal; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Open label single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Signos digital health app and CGM (Experimental): For all consented participants, the Signos app will use CGM data to provide recommendations customized to users for promoting general health and wellness.
  Interventions: Device: Continuous Glucose Monitor Device

INTERVENTIONS:
Device: Continuous Glucose Monitor Device — Continuous glucose monitoring automatically tracks blood glucose levels, also called blood sugar, throughout the day and night. You can see your glucose level anytime at a glance. You can also review how your glucose changes over a few hours or days to see trends. Seeing glucose levels in real time can help you make more informed decisions throughout the day about how to balance your food and physical activity.
  Other Names: CGM

SUMMARY:
Metabolic syndrome and resulting downstream health effects remains a growing health concern. In published trials, the use of continuous glucose monitoring (CGM) assists behavioral changes efforts, leading to improved adherence and results from diet and exercise changes in individuals with obesity, pre-diabetes and diabetes. Mobile health (mHealth) platforms provide satisfactory, easy-to-use tools that help participants in the pursuit of weight change goals. We hypothesize that the use of CGM data and targeted coaching and nutrition education will assist with weight optimization goals in the general (non-diabetic) population using the Signos mHealth platform, with associated health benefits.

DETAILED DESCRIPTION:
The scope of this study is to enroll existing and new Signos users in a volunteer study that utilizes a continuous glucose monitor (CGM) and mobile health application [Signos] to optimize general wellness and body weight and composition. This is a no more than minimal risk study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Own a smartphone and be willing to install the Signos App to use the app, receive messages or notifications, and input weight and other data.
* Willingness to complete questionaries or other surveys
* Able to speak and read English

Exclusion Criteria:

* Medical diagnosis of Type 1 Diabetes
* Medical diagnosis of Type 2 Diabetes
* Current medical diagnosis of an eating disorder (anorexia or bulimia) or previously struggled with disordered eating behaviors with current BMI less than 24
* Medical conditions (e.g., such as seizure disorder) requiring a specific medical diet.
* Inborn errors of metabolism such as phenylketonuria (PKU), glycogen storage disease, fructose intolerance, Maple Sugar Urine Disease (MSUD).
* Chronic or severe disease (e.g, chronic obstructive pulmonary disease [COPD], coronary artery disease, cerebrovascular accident [CVA], or cardiac arrhythmia) that would preclude a subject from safely participating in dietary recommendations and/or physical activity
* History of Gastric bypass or other bariatric surgery
* History of 10 or more soft tissue skin infections (such as cellulitis or abscesses)
* Intolerable skin reaction from adhesive
* Currently taking any of the following medications: Hydroxyurea, insulin, sulfonylureas, or medications prescribed specifically for the treatment of diagnosed diabetes
* Vulnerable populations such as minors, prisoners, or pregnant women will not be enrolled in this study. Women who become pregnant will be excluded at that time.
* Inability or unwillingness of subject to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31187 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Average fasting glucose | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  Daily fasting glucose, averaged periodically
Change in weight | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  Change in number of pounds

SECONDARY OUTCOMES:
Body composition | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  User input data including percentage of body fat or other measurements of body composition
Time in range | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  percentage of time spent "in range" glucose level less than 140 or as determined by other parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Signos, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall H, Perelman D, Breschi A, Limcaoco P, Kellogg R, McLaughlin T, Snyder M. Glucotypes reveal new patterns of glucose dysregulation. PLoS Biol. 2018 Jul 24;16(7):e2005143. doi: 10.1371/journal.pbio.2005143. eCollection 2018 Jul. PMID 30040822
- [Background] Adams OP. The impact of brief high-intensity exercise on blood glucose levels. Diabetes Metab Syndr Obes. 2013;6:113-22. doi: 10.2147/DMSO.S29222. Epub 2013 Feb 27. PMID 23467903
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Baron AD. Impaired glucose tolerance as a disease. Am J Cardiol. 2001 Sep 20;88(6A):16H-9H. doi: 10.1016/s0002-9149(01)01832-x. PMID 11576521
- [Background] Brown A, McArdle P, Taplin J, Unwin D, Unwin J, Deakin T, Wheatley S, Murdoch C, Malhotra A, Mellor D. Dietary strategies for remission of type 2 diabetes: A narrative review. J Hum Nutr Diet. 2022 Feb;35(1):165-178. doi: 10.1111/jhn.12938. Epub 2021 Sep 1. PMID 34323335
- [Background] Chin SO, Keum C, Woo J, Park J, Choi HJ, Woo JT, Rhee SY. Successful weight reduction and maintenance by using a smartphone application in those with overweight and obesity. Sci Rep. 2016 Nov 7;6:34563. doi: 10.1038/srep34563. PMID 27819345
- [Background] Ebbeling CB, Knapp A, Johnson A, Wong JMW, Greco KF, Ma C, Mora S, Ludwig DS. Effects of a low-carbohydrate diet on insulin-resistant dyslipoproteinemia-a randomized controlled feeding trial. Am J Clin Nutr. 2022 Jan 11;115(1):154-162. doi: 10.1093/ajcn/nqab287. PMID 34582545
- [Background] Ehrhardt N, Al Zaghal E. Behavior Modification in Prediabetes and Diabetes: Potential Use of Real-Time Continuous Glucose Monitoring. J Diabetes Sci Technol. 2019 Mar;13(2):271-275. doi: 10.1177/1932296818790994. Epub 2018 Aug 1. PMID 30066574
- [Background] The Lancet Diabetes Endocrinology. Metabolic health: a priority for the post-pandemic era. Lancet Diabetes Endocrinol. 2021 Apr;9(4):189. doi: 10.1016/S2213-8587(21)00058-9. Epub 2021 Mar 4. No abstract available. PMID 33676599
- [Background] Galderisi A, Giannini C, Weiss R, Kim G, Shabanova V, Santoro N, Pierpont B, Savoye M, Caprio S. Trajectories of changes in glucose tolerance in a multiethnic cohort of obese youths: an observational prospective analysis. Lancet Child Adolesc Health. 2018 Oct;2(10):726-735. doi: 10.1016/S2352-4642(18)30235-9. Epub 2018 Aug 24. PMID 30236381
- [Background] Gonzalez-Rodriguez M, Pazos-Couselo M, Garcia-Lopez JM, Rodriguez-Segade S, Rodriguez-Garcia J, Tunez-Bastida C, Gude F. Postprandial glycemic response in a non-diabetic adult population: the effect of nutrients is different between men and women. Nutr Metab (Lond). 2019 Jul 17;16:46. doi: 10.1186/s12986-019-0368-1. eCollection 2019. PMID 31346341
- [Background] Guyenet SJ, Schwartz MW. Clinical review: Regulation of food intake, energy balance, and body fat mass: implications for the pathogenesis and treatment of obesity. J Clin Endocrinol Metab. 2012 Mar;97(3):745-55. doi: 10.1210/jc.2011-2525. Epub 2012 Jan 11. PMID 22238401
- [Background] Hamley S, Kloosterman D, Duthie T, Dalla Man C, Visentin R, Mason SA, Ang T, Selathurai A, Kaur G, Morales-Scholz MG, Howlett KF, Kowalski GM, Shaw CS, Bruce CR. Mechanisms of hyperinsulinaemia in apparently healthy non-obese young adults: role of insulin secretion, clearance and action and associations with plasma amino acids. Diabetologia. 2019 Dec;62(12):2310-2324. doi: 10.1007/s00125-019-04990-y. Epub 2019 Sep 6. PMID 31489455
- [Background] Hyde PN, Sapper TN, Crabtree CD, LaFountain RA, Bowling ML, Buga A, Fell B, McSwiney FT, Dickerson RM, Miller VJ, Scandling D, Simonetti OP, Phinney SD, Kraemer WJ, King SA, Krauss RM, Volek JS. Dietary carbohydrate restriction improves metabolic syndrome independent of weight loss. JCI Insight. 2019 Jun 20;4(12):e128308. doi: 10.1172/jci.insight.128308. eCollection 2019 Jun 20. PMID 31217353
- [Background] Jagannathan R, Sevick MA, Fink D, Dankner R, Chetrit A, Roth J, Buysschaert M, Bergman M. The 1-hour post-load glucose level is more effective than HbA1c for screening dysglycemia. Acta Diabetol. 2016 Aug;53(4):543-50. doi: 10.1007/s00592-015-0829-6. Epub 2016 Jan 21. PMID 26794497
- [Background] Jakubowicz D, Barnea M, Wainstein J, Froy O. High caloric intake at breakfast vs. dinner differentially influences weight loss of overweight and obese women. Obesity (Silver Spring). 2013 Dec;21(12):2504-12. doi: 10.1002/oby.20460. Epub 2013 Jul 2. PMID 23512957
- [Background] Ludwig DS, Aronne LJ, Astrup A, de Cabo R, Cantley LC, Friedman MI, Heymsfield SB, Johnson JD, King JC, Krauss RM, Lieberman DE, Taubes G, Volek JS, Westman EC, Willett WC, Yancy WS, Ebbeling CB. The carbohydrate-insulin model: a physiological perspective on the obesity pandemic. Am J Clin Nutr. 2021 Dec 1;114(6):1873-1885. doi: 10.1093/ajcn/nqab270. PMID 34515299
- [Background] Di Flaviani A, Picconi F, Di Stefano P, Giordani I, Malandrucco I, Maggio P, Palazzo P, Sgreccia F, Peraldo C, Farina F, Frajese G, Frontoni S. Impact of glycemic and blood pressure variability on surrogate measures of cardiovascular outcomes in type 2 diabetic patients. Diabetes Care. 2011 Jul;34(7):1605-9. doi: 10.2337/dc11-0034. Epub 2011 May 24. PMID 21610126
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Brynes AE, Adamson J, Dornhorst A, Frost GS. The beneficial effect of a diet with low glycaemic index on 24 h glucose profiles in healthy young people as assessed by continuous glucose monitoring. Br J Nutr. 2005 Feb;93(2):179-82. doi: 10.1079/bjn20041318. PMID 15788110
- [Background] Liao Y, Schembre S. Acceptability of Continuous Glucose Monitoring in Free-Living Healthy Individuals: Implications for the Use of Wearable Biosensors in Diet and Physical Activity Research. JMIR Mhealth Uhealth. 2018 Oct 24;6(10):e11181. doi: 10.2196/11181. PMID 30355561
- [Background] Neri D, Martinez-Steele E, Monteiro CA, Levy RB. Consumption of ultra-processed foods and its association with added sugar content in the diets of US children, NHANES 2009-2014. Pediatr Obes. 2019 Dec;14(12):e12563. doi: 10.1111/ijpo.12563. Epub 2019 Jul 30. PMID 31364315
- [Background] Page KA, Seo D, Belfort-DeAguiar R, Lacadie C, Dzuira J, Naik S, Amarnath S, Constable RT, Sherwin RS, Sinha R. Circulating glucose levels modulate neural control of desire for high-calorie foods in humans. J Clin Invest. 2011 Oct;121(10):4161-9. doi: 10.1172/JCI57873. Epub 2011 Sep 19. PMID 21926468
- [Background] Painter SL, Lu W, Schneider J, James R, Shah B. Drivers of weight loss in a CDC-recognized digital diabetes prevention program. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001132. doi: 10.1136/bmjdrc-2019-001132. PMID 32624481
- [Background] Suh S, Kim JH. Glycemic Variability: How Do We Measure It and Why Is It Important? Diabetes Metab J. 2015 Aug;39(4):273-82. doi: 10.4093/dmj.2015.39.4.273. PMID 26301188
- [Background] Turk MW, Elci OU, Wang J, Sereika SM, Ewing LJ, Acharya SD, Glanz K, Burke LE. Self-monitoring as a mediator of weight loss in the SMART randomized clinical trial. Int J Behav Med. 2013 Dec;20(4):556-61. doi: 10.1007/s12529-012-9259-9. PMID 22936524
- [Background] Wang Y, Xue H, Huang Y, Huang L, Zhang D. A Systematic Review of Application and Effectiveness of mHealth Interventions for Obesity and Diabetes Treatment and Self-Management. Adv Nutr. 2017 May 15;8(3):449-462. doi: 10.3945/an.116.014100. Print 2017 May. PMID 28507010
- [Background] Wyatt P, Berry SE, Finlayson G, O'Driscoll R, Hadjigeorgiou G, Drew DA, Khatib HA, Nguyen LH, Linenberg I, Chan AT, Spector TD, Franks PW, Wolf J, Blundell J, Valdes AM. Postprandial glycaemic dips predict appetite and energy intake in healthy individuals. Nat Metab. 2021 Apr;3(4):523-529. doi: 10.1038/s42255-021-00383-x. Epub 2021 Apr 12. PMID 33846643
- [Background] Yang X, Zhu Y, Luo S, Chen L, Yan J, Zeng L, Xu W, Weng J. [Glucose characteristics in normal glucose tolerance subjects with metabolic syndrome]. Zhonghua Yi Xue Za Zhi. 2015 Apr 14;95(14):1070-3. Chinese. PMID 26081206
- [Background] Allen NA, Fain JA, Braun B, Chipkin SR. Continuous glucose monitoring counseling improves physical activity behaviors of individuals with type 2 diabetes: A randomized clinical trial. Diabetes Res Clin Pract. 2008 Jun;80(3):371-9. doi: 10.1016/j.diabres.2008.01.006. Epub 2008 Mar 4. PMID 18304674
- [Background] Azami Y, Funakoshi M, Matsumoto H, Ikota A, Ito K, Okimoto H, Shimizu N, Tsujimura F, Fukuda H, Miyagi C, Osawa S, Osawa R, Miura J. Long working hours and skipping breakfast concomitant with late evening meals are associated with suboptimal glycemic control among young male Japanese patients with type 2 diabetes. J Diabetes Investig. 2019 Jan;10(1):73-83. doi: 10.1111/jdi.12852. Epub 2018 May 30. PMID 29667372
- [Background] Bailey KJ, Little JP, Jung ME. Self-Monitoring Using Continuous Glucose Monitors with Real-Time Feedback Improves Exercise Adherence in Individuals with Impaired Blood Glucose: A Pilot Study. Diabetes Technol Ther. 2016 Mar;18(3):185-93. doi: 10.1089/dia.2015.0285. Epub 2016 Feb 17. PMID 26885934
- [Background] Cox DJ, Taylor AG, Moncrief M, Diamond A, Yancy WS Jr, Hegde S, McCall AL. Continuous Glucose Monitoring in the Self-management of Type 2 Diabetes: A Paradigm Shift. Diabetes Care. 2016 May;39(5):e71-3. doi: 10.2337/dc15-2836. Epub 2016 Mar 17. No abstract available. PMID 26989181
- [Background] Freckmann G, Hagenlocher S, Baumstark A, Jendrike N, Gillen RC, Rossner K, Haug C. Continuous glucose profiles in healthy subjects under everyday life conditions and after different meals. J Diabetes Sci Technol. 2007 Sep;1(5):695-703. doi: 10.1177/193229680700100513. PMID 19885137
- [Background] Hatamoto Y, Goya R, Yamada Y, Yoshimura E, Nishimura S, Higaki Y, Tanaka H. Effect of exercise timing on elevated postprandial glucose levels. J Appl Physiol (1985). 2017 Aug 1;123(2):278-284. doi: 10.1152/japplphysiol.00608.2016. Epub 2017 Apr 13. PMID 28408695
- [Background] Jakubowicz D, Wainstein J, Ahren B, Landau Z, Bar-Dayan Y, Froy O. Fasting until noon triggers increased postprandial hyperglycemia and impaired insulin response after lunch and dinner in individuals with type 2 diabetes: a randomized clinical trial. Diabetes Care. 2015 Oct;38(10):1820-6. doi: 10.2337/dc15-0761. Epub 2015 Jul 28. PMID 26220945
- [Background] Juanola-Falgarona M, Salas-Salvado J, Ibarrola-Jurado N, Rabassa-Soler A, Diaz-Lopez A, Guasch-Ferre M, Hernandez-Alonso P, Balanza R, Bullo M. Effect of the glycemic index of the diet on weight loss, modulation of satiety, inflammation, and other metabolic risk factors: a randomized controlled trial. Am J Clin Nutr. 2014 Jul;100(1):27-35. doi: 10.3945/ajcn.113.081216. Epub 2014 Apr 30. PMID 24787494
- [Background] Kolb H, Stumvoll M, Kramer W, Kempf K, Martin S. Insulin translates unfavourable lifestyle into obesity. BMC Med. 2018 Dec 13;16(1):232. doi: 10.1186/s12916-018-1225-1. PMID 30541568
- [Background] Kong LC, Wuillemin PH, Bastard JP, Sokolovska N, Gougis S, Fellahi S, Darakhshan F, Bonnefont-Rousselot D, Bittar R, Dore J, Zucker JD, Clement K, Rizkalla S. Insulin resistance and inflammation predict kinetic body weight changes in response to dietary weight loss and maintenance in overweight and obese subjects by using a Bayesian network approach. Am J Clin Nutr. 2013 Dec;98(6):1385-94. doi: 10.3945/ajcn.113.058099. Epub 2013 Oct 30. PMID 24172304
- [Background] Rynders CA, Blanc S, DeJong N, Bessesen DH, Bergouignan A. Sedentary behaviour is a key determinant of metabolic inflexibility. J Physiol. 2018 Apr 15;596(8):1319-1330. doi: 10.1113/JP273282. Epub 2017 Jul 4. PMID 28543022
- [Background] Lin HJ, Lee BC, Ho YL, Lin YH, Chen CY, Hsu HC, Lin MS, Chien KL, Chen MF. Postprandial glucose improves the risk prediction of cardiovascular death beyond the metabolic syndrome in the nondiabetic population. Diabetes Care. 2009 Sep;32(9):1721-6. doi: 10.2337/dc08-2337. Epub 2009 Jun 5. PMID 19502543
- [Background] Shukla AP, Dickison M, Coughlin N, Karan A, Mauer E, Truong W, Casper A, Emiliano AB, Kumar RB, Saunders KH, Igel LI, Aronne LJ. The impact of food order on postprandial glycaemic excursions in prediabetes. Diabetes Obes Metab. 2019 Feb;21(2):377-381. doi: 10.1111/dom.13503. Epub 2018 Sep 10. PMID 30101510
- [Background] Soliman A, DeSanctis V, Yassin M, Elalaily R, Eldarsy NE. Continuous glucose monitoring system and new era of early diagnosis of diabetes in high risk groups. Indian J Endocrinol Metab. 2014 May;18(3):274-82. doi: 10.4103/2230-8210.131130. PMID 24944918
- [Background] Velasquez-Mieyer PA, Cowan PA, Arheart KL, Buffington CK, Spencer KA, Connelly BE, Cowan GW, Lustig RH. Suppression of insulin secretion is associated with weight loss and altered macronutrient intake and preference in a subset of obese adults. Int J Obes Relat Metab Disord. 2003 Feb;27(2):219-26. doi: 10.1038/sj.ijo.802227. PMID 12587002
- [Background] Yoo HJ, An HG, Park SY, Ryu OH, Kim HY, Seo JA, Hong EG, Shin DH, Kim YH, Kim SG, Choi KM, Park IB, Yu JM, Baik SH. Use of a real time continuous glucose monitoring system as a motivational device for poorly controlled type 2 diabetes. Diabetes Res Clin Pract. 2008 Oct;82(1):73-9. doi: 10.1016/j.diabres.2008.06.015. Epub 2008 Aug 12. PMID 18701183
- [Background] Haxhi J, Scotto di Palumbo A, Sacchetti M. Exercising for metabolic control: is timing important? Ann Nutr Metab. 2013;62(1):14-25. doi: 10.1159/000343788. Epub 2012 Nov 27. PMID 23208206
- [Background] Kim J, Lam W, Wang Q, Parikh L, Elshafie A, Sanchez-Rangel E, Schmidt C, Li F, Hwang J, Belfort-DeAguiar R. In a Free-Living Setting, Obesity Is Associated With Greater Food Intake in Response to a Similar Premeal Glucose Nadir. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3911-3919. doi: 10.1210/jc.2019-00240. PMID 31087061
- [Background] Mendes-Soares H, Raveh-Sadka T, Azulay S, Edens K, Ben-Shlomo Y, Cohen Y, Ofek T, Bachrach D, Stevens J, Colibaseanu D, Segal L, Kashyap P, Nelson H. Assessment of a Personalized Approach to Predicting Postprandial Glycemic Responses to Food Among Individuals Without Diabetes. JAMA Netw Open. 2019 Feb 1;2(2):e188102. doi: 10.1001/jamanetworkopen.2018.8102. PMID 30735238
- [Background] Penckofer S, Quinn L, Byrn M, Ferrans C, Miller M, Strange P. Does glycemic variability impact mood and quality of life? Diabetes Technol Ther. 2012 Apr;14(4):303-10. doi: 10.1089/dia.2011.0191. Epub 2012 Feb 10. PMID 22324383
- [Background] Steinberg DM, Bennett GG, Askew S, Tate DF. Weighing every day matters: daily weighing improves weight loss and adoption of weight control behaviors. J Acad Nutr Diet. 2015 Apr;115(4):511-8. doi: 10.1016/j.jand.2014.12.011. Epub 2015 Feb 12. PMID 25683820
- [Background] Chandler-Laney PC, Morrison SA, Goree LL, Ellis AC, Casazza K, Desmond R, Gower BA. Return of hunger following a relatively high carbohydrate breakfast is associated with earlier recorded glucose peak and nadir. Appetite. 2014 Sep;80:236-41. doi: 10.1016/j.appet.2014.04.031. Epub 2014 May 10. PMID 24819342